CLINICAL TRIAL: NCT00003270
Title: Cord Blood Transplantation for Hematologic Malignancies and Bone Marrow Failure Syndromes
Brief Title: Chemotherapy, Radiation Therapy, and Umbilical Cord Blood Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS 97-26; DS 97-26
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; Burkitt lymphoma; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent/refractory childhood Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; graft versus host disease; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Burkitt Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Antilymphocyte Serum; Filgrastim; Busulfan; Cyclophosphamide; Cyclosporine; Methylprednisolone; Cord Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Patients eligible to undergo total body irradiation (TBI) first receive cyclophosphamide IV over 2 hours on days -5 and -4, then undergo TBI twice a day on days -3 to -1. Patients also receive antithymocyte globulin (ATG) IV over 10 hours on days -3 to -1. Cord blood is infused on day 0
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Drug: busulfan; Drug: cyclophosphamide; Drug: cyclosporine; Drug: methylprednisolone; Procedure: bone marrow ablation with stem cell support; Procedure: umbilical cord blood transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: anti-thymocyte globulin — IV
Biological: filgrastim — IV
Drug: busulfan — IV
Drug: cyclophosphamide — IV
Drug: cyclosporine — IV
Drug: methylprednisolone — IV
Procedure: bone marrow ablation with stem cell support — IV
Procedure: umbilical cord blood transplantation — IV
Radiation: radiation therapy — High energy X-rays

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Umbilical cord blood transplantation may allow doctors to give higher doses of chemotherapy or radiation therapy and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy, radiation therapy, and umbilical cord blood transplantation in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety, efficacy, and toxicity of using cord blood as a source for stem cell transplantation in patients with hematologic malignancies.

OUTLINE: Patients undergo autologous bone marrow harvesting or peripheral stem cell collection prior to transplant regimen, unless the patient has acute leukemia in relapse, aplastic anemia, or myelodysplastic syndrome. Arm I: Patients eligible to undergo total body irradiation (TBI) first receive cyclophosphamide IV over 2 hours on days -5 and -4, then undergo TBI twice a day on days -3 to -1. Patients also receive antithymocyte globulin (ATG) IV over 10 hours on days -3 to -1. Cord blood is infused on day 0. Arm II: Patients not eligible to receive TBI receive oral busulfan every 6 hours on days -7 to -4 for a total of 16 doses. Cyclophosphamide, ATG, and cord blood are then administered as in arm I. All patients receive cyclosporine on days -2 to 180, methylprednisolone on days 5-180, and filgrastim (G-CSF) from day 1. Patients are followed weekly until day 180 and then monthly for 2 years.

PROJECTED ACCRUAL: A total of 20 patients (10 patients per arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven hematologic malignancy Acute lymphocytic leukemia (ALL): In second or later remission In first remission with poor prognostic features (Philadelphia chromosome positive) Acute myeloid leukemia (AML): In second or later remission In first remission with poor prognostic features, e.g., Arising from myelodysplastic syndrome Cytogenetics with -5, -7, +8, 11q23 abnormalities Complex cytogenetics AML or ALL refractory to induction or in relapse Myelodysplastic syndrome Chronic myelogenous leukemia Severe aplastic anemia or Fanconi's anemia Relapsed Hodgkin's disease Relapsed non-Hodgkin's lymphoma Multiple myeloma No suitable family donor matched for 5 or 6 HLA antigens (A, B, DR) No suitable unrelated donor matched for 6 HLA antigens Cord blood donor available matched for 4-6 out of 6 HLA antigens

PATIENT CHARACTERISTICS: Age: 5 to 50 Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 3 times normal Alkaline phosphatase less than 3 times normal SGOT less than 3 times normal Renal: Creatinine less than 2 times normal OR Creatinine clearance greater than 60 mL/min Cardiovascular: MUGA with ejection fraction at least 50% Pulmonary: DLCO and spirometry at least 60% OR Exercise VO2 max/kg at least 15 mL/min/kg Other: HIV antibody negative Hepatitis B surface antigen negative No active bacterial, viral, or fungal infection

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy allowed If following limits have not been exceeded, patient may receive total body irradiation: No prior radiation to one entire kidney Whole liver received no greater than 1000 cGy No prior whole abdomen radiotherapy Small bowel received no greater than 3000 cGy Heart received no greater than 1800 cGy No prior whole lung radiotherapy CNS received less than 30 cGy (whole brain or any portion of the spine) Surgery: Not specified

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 1997-09-04 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Jean Bambach, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Eligible patients are treated with busulfan IV over 2 hours on days -7 to -4, cyclophosphamide IV over 2 hours on days -3 and -2, antithymocyte globulin (ATG) IV over 10 hours on days -3 to -1 (BuCyATG) and cord blood is infused on day 0; or are treated with cyclophosphamide IV over 2 hours on days -5 and -4, antithymocyte globulin (ATG) IV over 10 hours on days -3 to -1, and undergo TBI twice a day on days -3 to -1 (CyATGTBI) and cord blood is infused on day 0
Period: Overall Study
Arm/Group | Arm 1
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 32.5 [5 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Disease [Count of Participants; unit: Participants]
  ALL | 3
  AML | 5
  Aplastic Anemia | 1
  CML | 7
  MDS/MPD | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Continuous complete remission (for patients in complete remission before treatment) or induced complete remission (for patients not in complete remission before treatment)
Time Frame: day +100 after Cord Blood Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 20
Participants
  CR/CCR | 12
  Progressed | 1
  Not evaluable (early death) | 7

2. Secondary Outcome: Progression-free Survival
Description: time to disease progression or death due to any cause
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 20
% of participants | 50 [28 to 72]

ADVERSE EVENTS:
Time Frame: Adverse Event, Serious Adverse Event and All Cause Mortality are from start of treatment (Day -7 or -5) through day +100 after cord blood infusion
Description: SAE is delayed engraftment or failed to engraft Died before engraftment is defined as death before Absolute Neutrophil Count recovery Failure to engraft is defined as survival until at least day +42 without Absolute Neutrophil Count recovery Other AEs include acute GVHD grade III-IV and RRT grade 3-4 RRT is defined using Bearman Regimen Related Toxicity Criteria Acute GVHD grade III-IV is defined using Glucksberg criteria
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 8/20
Serious Adverse Events (participants affected / at risk) | 5/20
Other Adverse Events (participants affected / at risk) | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=20)
DBE/FTE (Blood and lymphatic system disorders) | 5 (5) — DBE: Died before engraftment (did not achieve absolute neutrophil recovery) FTE: Failed to engraft (survived to at least day +42 without absolute neutrophil recovery
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=20)
Severe Acute graft-versus-host disease (Immune system disorders) | 5 (5) — Overall grade III-IV acute graft-versus-host disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT00003270/Prot_SAP_000.pdf